CLINICAL TRIAL: NCT04024540
Title: Isocaloric Dietary Restriction vs. Bariatric Surgery for Obesity Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wang Weiqing, professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ruijin-2019-34
Record Dates: First submitted 2019-07-13; First posted 2019-07-18 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- isocaloric dietary restriction (Experimental): Very low caloric diet 400 kcal/d for a week, 600 kcal/d for another week and 800 kcal/d for 2 weeks.
  Interventions: Dietary Supplement: isocaloric dietary restriction
- Bariatric surgery (Active Comparator): Laparoscopic vertical sleeve gastrectomy
  Interventions: Dietary Supplement: isocaloric dietary restriction; Procedure: Bariatric surgery

INTERVENTIONS:
Dietary Supplement: isocaloric dietary restriction — Very low caloric diet
Procedure: Bariatric surgery — Laparoscopic vertical sleeve gastrectomy
  Arms: Bariatric surgery

SUMMARY:
This is a prospective, randomized, two-armed study to assess the efficacy and safety of isocaloric dietary restriction in the treatment of obese without diabetic for a period of 4 weeks.

DETAILED DESCRIPTION:
This is a randomized, open-label, two arms trial. Based on inclusion and exclusion criteria, 72 eligible patients, who are 18-45 years old, with BMI between 35 to 45kg/m2 are assigned to one of two intervention groups: isocaloric dietary restriction; bariatric surgery. Both groups were given a dietary intervention for a period of 4 weeks (in rigorous supervision confined in inpatient department). The main purpose of this study is to clarify the efficacy of isocaloric dietary restriction, compared to bariatric surgery, in losing weight and improving metabolic factors. This is an investigator-initiated study performed by department of endocrinology and metabolic disease, Ruijin hospital affiliated with Shanghai Jiaotong University School of Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 45 years old
* 35 ≤ BMI ≤ 45 kg/m2

Exclusion Criteria:

* Obesity induced by other endocrinologic disorders
* Severe gastrointestinal diseases or contraindication for surgery
* History or newly known of diabetes
* Use of hypoglycemic medications, antibiotic in the preceding 2 months, or yogurt within 5 days
* Weight change more than 5% of body weight within the past 3 months
* Severe or unstable cardiovascular, liver or renal diseases or known cancer
* History of drug or alcohol abuse or other substance abuse
* Any mental disorders or current use of antidepressantsPregnancy or lactation or consideration of pregnancy
* Allergies to specific food ingredients in the intervention

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Body weight | 4 weeks
  Change of body weight (kg) from baseline measured by study personnel.

SECONDARY OUTCOMES:
Body mass index | 4 weeks
  Change of BMI [BMI = weight (kg)/height2(m2)] from baseline measured by study personnel.
Waist, hip and neck circumference | 4 weeks
  Waist, hip and neck circumference (cm) measured by study personnel.
Body composition | 4 weeks
  Body fat mass, fat free mass (kg) and body fat rate measured by DEXA.
Liver fat content | 4 weeks
  Liver fat content measured by MRI.
Energy expenditure | 4 weeks
  Energy expenditure measured by metabolic chamber.
Glucose metabolism | 4 weeks
  including glycated haemoglobin, HOMA-IR, fasting plasma glucose levels and serum insulin levels, post-prandial plasma glucose levels and serum insulin levels (using mixed-meal test).
Lipid profiles | 4 weeks
  including serum triglycerides, total cholesterol, low-density lipoproteins cholesterol and high-density lipoproteins cholesterol.
Gut hormones | 4 weeks
  including Glucagon-like peptide 1, gastric inhibitory polypeptide, ghrelin, peptide YY and etc.
Hepatic function | 4 weeks
  including alanine aminotransferase, aspartate aminotransferase, γ-glutamyltransferase, and alkaline phosphatase.
Renal function | 4 weeks
  including serum urea nitrogen, serum creatinine, and serum urinary acid.
Endocrine hormones | 4 weeks
  including thyroid function, sex hormone, insulin-like growth factor and etc.
Appetite (the subjective desire to eat) | 4 weeks
  assessed according to TFEQ-R21
Adverse events | 4 weeks
  Safety outcomes
Systolic and diastolic blood pressure | 4 weeks
  Safety outcomes
Body temperature | 4 weeks
  Safety outcomes
Pulse rate | 4 weeks
  Safety outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Weiqing Wang, M.D. Ph.D., Principal Investigator — Shanghai Clinic Center for Endocrine and Metabolic Diseases, Ruijin Hospital, Shanghai Institute for Endocrine and Metabolic Diseases
Locations (1):
- Ruijin hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China